CLINICAL TRIAL: NCT06338176
Title: Optimizing the Management of Staphylococcus Aureus Bacteremia (OPTIMUS-SAB): A Stepped Wedge Clinical Trial Evaluating the Effectiveness of a Centralized S. Aureus Management Model
Brief Title: Optimizing the Management of Staphylococcus Aureus Bacteremia (OPTIMUS-SAB)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alberta (Other)
Collaborators: Alberta Health services (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: Pro00128904
Record Dates: First submitted 2024-03-23; First posted 2024-03-29 (Actual); Last update posted 2025-07-08 (Actual); Status verified 2025-07

CONDITIONS: Staph Aureus Bacteremia
Keywords: care pathway; infectious disease consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OPTIMUS-SAB care pathway (Experimental): Province-wide real time automated notifications of new SAB cases will be established and delivered to a centralized SAB care team electronically through Connect Care. The centralized SAB care team consists of a SAB clinical coordinator, ID specialists and other ad hoc representation depending on patient needs. Following patient chart review, the centralized SAB care team contacts the most responsible physician (MRP) to provide preliminary recommendations to optimize care, both verbally and in written format, facilitated by Connect Care (Alberta Health Services electronic medical record).
  Interventions: Other: OPTIMUS-SAB clinical care pathway
- Standard of care (No Intervention)

INTERVENTIONS:
Other: OPTIMUS-SAB clinical care pathway — Activation of SAB clinical care pathway within EMR system.
  Arms: OPTIMUS-SAB care pathway

SUMMARY:
Staphylococcus aureus bacteremia (SAB) is associated with high morbidity and mortality rates with an incidence disproportionately higher in vulnerable populations. Management according to evidence-based care parameters, in particular Infectious Diseases (ID) consultation, is associated with improved mortality. SAB management is suboptimal in Alberta compared to other jurisdictions. An Alberta-based pilot study confirmed that timely recommendations to optimize SAB care, including ID consultation, was associated with improved adherence to all evidence-based quality-of-care indicators.

Leveraging this pilot work, the investigators aim to implement OPTIMUS-SAB, an enhanced model of the pilot, to optimize and standardize SAB management across Alberta. The implementation study will be a zone-based acute care site stepped wedge design. OPTIMUS-SAB will consist of a centralized SAB care team whom will receive automated notification of all blood cultures positive for S. aureus allowing them to review the patient's medical chart and make preliminary management recommendations according to an evidence-based care bundle.

The investigators will evaluate adherence to evidence-based SAB quality-of-care indicators before and after OPTIMUS-SAB implementation and expect this to improve with a resultant reduction in duration of bacteremia, length of stay, readmission rates, and mortality. In turn, this will translate into cost savings for the health care system.

ELIGIBILITY:
Inclusion Criteria:

* Age greater than 18 years at the time of hospital admission
* Confirmed S. aureus bacteremia by blood culture performed at a laboratory in Alberta, Canada
* Admitted to a designated acute care site in Alberta, Canada

Exclusion Criteria:

* The treating team believes death is imminent or inevitable .
* GCD are C-level within 48 hours of admission.
* The patient is transferred in from an out-of-province acute care center with a pre-existing SAB diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1800 (Estimated)
Dates: Start 2024-05-01 (Actual); Primary Completion 2025-10-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Adherence to quality-of-care indicators | Within 90 days
  Defined as:
  1. ID involvement and time to ID involvement, defined by the presence of an ID consult note and/or recommendations in the chart.
  2. Repeat blood cultures, to document clearance of bacteremia, within 72 hours from the last positive blood culture.
  3. Guideline-concordant empiric antibiotic administered and time to receipt.
  4. Guideline concordant definitive antibiotic administered and time to receipt.
  5. Therapeutic drug monitoring of patents treatments with vancomycin.
  6. Appropriate dose adjustment of antimicrobials based on renal function according to local guidelines.
  7. Echocardiogram (transthoracic or transesophageal) performed within 72 hours of diagnosis.
  8. Source control achieved.
  9. Appropriate duration of antibiotic therapy ordered and delivered.

SECONDARY OUTCOMES:
Length of stay | 180 days maximum
  Acute hospital length of stay
Hospital re-admission rates | 90 days
  re-admission to acute care rate
All-cause mortality | 180 days
  death from any cause
In hospital mortality | 90 days
  death within hospital stay
Costing evaluation | One year
  Cost of SAB treatment related to hospitalization, including physician provision of care, and antibiotics.
Implementation evaluation | 3 years
  User experience and feedback from patients and providers will be collected at the start and end of each active implementation phase. This information will be paired with assessments of barriers, facilitators, and contextual factors informed by the Consolidated Framework for Implementation Research (CFIR) and Normalization Process Theory during the pre-implementation phase and at the end of active implementation.

CONTACTS AND LOCATIONS:
Overall Officials: Justin Chen, MD, Principal Investigator — University of Alberta
Locations (101):
- Canada (101):
  - Athabasca Healthcare Centre, Athabasca, Alberta
  - Mineral Springs Hospital, Banff, Alberta
  - Barrhead Healthcare Centre, Barrhead, Alberta
  - Bassano Health Centre, Bassano, Alberta
  - Beaverlodge Municipal Hospital, Beaverlodge, Alberta
  - Oilfields General Hospital, Black Diamond, Alberta
  - Bonnyville Healthcare Centre, Bonnyville, Alberta
  - Bow Island Health Centre, Bow Island, Alberta
  - Boyle Healthcare Centre, Boyle, Alberta
  - Brooks Health Centre, Brooks, Alberta
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Foothills Medical Centre, Calgary, Alberta
  - Peter Lougheed Centre, Calgary, Alberta
  - South Health Campus, Calgary, Alberta
  - Tom Baker Cancer Centre, Calgary, Alberta
  - St. Mary's Hospital, Camrose, Alberta
  - Canmore General Hospital, Canmore, Alberta
  - Cardston Health Centre, Cardston, Alberta
  - Our Lady of the Rosary Hospital, Castor, Alberta
  - Claresholm General Hospital, Claresholm, Alberta
  - Coaldale Health Centre, Coaldale, Alberta
  - Cold Lake Healthcare Centre, Cold Lake, Alberta
  - Consort Hospital and Care Centre, Consort, Alberta
  - Coronation Hospital and Care Centre, Coronation, Alberta
  - Crowsnest Pass Health Centre, Crowsnest Pass, Alberta
  - Daysland Health Centre, Daysland, Alberta
  - Devon General Hospital, Devon, Alberta
  - Didsbury District Health Services, Didsbury, Alberta
  - Drayton Valley Hospital and Care Centre, Drayton Valley, Alberta
  - Drumheller Health Centre, Drumheller, Alberta
  - Cross Cancer Institute, Edmonton, Alberta
  - Glenrose Rehabilitation Hospital, Edmonton, Alberta
  - Grey Nuns Community Hospital, Edmonton, Alberta
  - Misericordia Community Hospital, Edmonton, Alberta
  - Royal Alexandra Hospital, Edmonton, Alberta
  - University of Alberta Hospital, Edmonton, Alberta
  - Edson Healthcare Centre, Edson, Alberta
  - Elk Point Healthcare Centre, Elk Point, Alberta
  - Fairview Health Complex, Fairview, Alberta
  - Northern Lights Regional Health Centre, Fort McMurray, Alberta
  - St. Theresa General Hospital, Fort Vermilion, Alberta
  - Fox Creek Healthcare Centre, Fox Creek, Alberta
  - Fort Saskatchewan Community Hospital, Ft Saskatchewan, Alberta
  - Grande Cache Community Health Complex, Grande Cache, Alberta
  - Grande Prairie Regional Hospital, Grande Prairie, Alberta
  - Grimshaw / Berwyn and District Community Health Centre, Grimshaw, Alberta
  - Hanna Health Centre, Hanna, Alberta
  - Hardisty Health Centre, Hardisty, Alberta
  - Northwest Health Centre, High Level, Alberta
  - High Prairie Health Complex, High Prairie, Alberta
  - High River General Hospital, High River, Alberta
  - Hinton Healthcare Centre, Hinton, Alberta
  - Innisfail Health Centre, Innisfail, Alberta
  - Seton - Jasper Healthcare Centre, Jasper, Alberta
  - Killam Health Centre, Killam, Alberta
  - William J Cadzow - Lac La Biche Health Care Centre, Lac La Biche, Alberta
  - Lacombe Hospital, Lacombe, Alberta
  - Lamont Health Centre, Lamont, Alberta
  - Leduc Community Hospital, Leduc, Alberta
  - Chinook Regional Hospital, Lethbridge, Alberta
  - Lloydminster Hospital, Lloydminster, Alberta
  - Manning Community Health Centre, Manning, Alberta
  - Mayerthorpe Healthcare Centre, Mayerthorpe, Alberta
  - Sacred Heart Community Healt, McLennan, Alberta
  - Medicine Hat Regional Hospital, Medicine Hat, Alberta
  - Olds Hospital and Care Centre, Olds, Alberta
  - Big Country Hospital, Oyen, Alberta
  - Peace River Community Health Centre, Peace River, Alberta
  - Pincher Creek Health Centre, Pincher Creek, Alberta
  - Ponoka Hospital, Ponoka, Alberta
  - Provost Health Centre, Provost, Alberta
  - Raymond Health Centre, Raymond, Alberta
  - Red Deer Regional Hospital Centre, Red Deer, Alberta
  - Redwater Health Centre, Redwater, Alberta
  - Rimbey Hospital, Rimbey, Alberta
  - Rocky Mountain House Health Centre, Rocky Mountain House, Alberta
  - Rockyview General Hospital, Rockyview, Alberta
  - Slave Lake Healthcare Centre, Slave Lake, Alberta
  - George McDougall - Smoky Lake Healthcare Centre, Smoky Lake, Alberta
  - Central Peace Health Complex, Spirit River, Alberta
  - Sturgeon Community Hospital, St. Albert, Alberta
  - St. Therese - St. Paul Healthcare Centre, St. Paul, Alberta
  - Stettler Hospital, Stettler, Alberta
  - Strathmore District Health Services, Strathmore, Alberta
  - Myron Thompson Health Centre, Sundre, Alberta
  - Swan Hills Healthcare Centre, Swan Hills, Alberta
  - Taber Health Centre, Taber, Alberta
  - Three Hills Health Centre, Three Hills, Alberta
  - Tofield Health Centre, Tofield, Alberta
  - Two Hills Health Centre, Two Hills, Alberta
  - Valleyview Health Centre, Valleyview, Alberta
  - St. Joseph's General Hospital, Vegreville, Alberta
  - Vermilion Health Centre, Vermilion, Alberta
  - Viking Health Centre, Viking, Alberta
  - Vulcan Community Health Centre, Vulcan, Alberta
  - Wabasca/Desmarais Healthcare Centre, Wabasca, Alberta
  - Wainwright Health Centre, Wainwright, Alberta
  - Westlock Healthcare Centre, Westlock, Alberta
  - Westview Health Centre, Westview Village, Alberta
  - Wetaskiwin Hospital, Wetaskiwin, Alberta
  - Whitecourt Healthcare Centre, Whitecourt, Alberta

REFERENCES:
- [Background] Remtulla S, Zurek K, Cervera C, Hernandez C, Lee MC, Hoang HL. Impact of an Unsolicited, Standardized Form-Based Antimicrobial Stewardship Intervention to Improve Guideline Adherence in the Management of Staphylococcus aureus Bacteremia. Open Forum Infect Dis. 2019 Feb 26;6(4):ofz098. doi: 10.1093/ofid/ofz098. eCollection 2019 Apr. PMID 30949538